CLINICAL TRIAL: NCT03211013
Title: Placebo-Controlled Study of the Effects of Oxytocin on Attentional Bias and Startle in PTSD
Brief Title: Study of the Effects of Oxytocin on Attentional Bias and Startle in PTSD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Steven Woodward, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: WOS0022ADM
Record Dates: First submitted 2017-04-03; First posted 2017-07-07 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: oxytocin; PTSD; attention bias; startle
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized double-blind crossover design, in which all participants will undergo 2 sessions, receiving either oxytocin nasal spray or placebo nasal spray in random order.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding of oxytocin drug container + randomization of oxytocin/placebo ordering over sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immediate Oxytocin (Experimental): Participants randomly assigned to this arm will receive OT nasal spray (24 IU) at laboratory visit 1 and placebo nasal spray at visit 2. The order will be masked for participants and study staff.
  Interventions: Drug: Oxytocin; Drug: Placebos
- Delayed Oxytocin (Placebo Comparator): Participants randomly assigned to this arm will receive placebo nasal spray at laboratory visit 1 and OT nasal spray (24 IU) at visit 2. The order will be masked for participants and study staff.
  Interventions: Drug: Oxytocin; Drug: Placebos

INTERVENTIONS:
Drug: Oxytocin — single-dose administration of OT nasal spray, complete computer-based tasks post-dose for approximately 1 hour
  Other Names: syntocinon
Drug: Placebos — single-dose administration of placebo nasal spray, complete computer-based tasks post-dose for approximately 1 hour

SUMMARY:
The investigators will test whether intranasal oxytocin (24 IU vs placebo) will induce effects on attention bias and startle comparable to those the investigators have shown to be induced by the presence (vs absence) of a service dog in Veterans diagnosed with PTSD. This possibility is suggested by a 2015 study showing that urinary oxytocin levels are elevated in association with mutual gaze between dogs and their owners.

DETAILED DESCRIPTION:
Background and significance:

Chronic severe posttraumatic stress disorder (PTSD) is among the most prevalent and expensive diagnoses addressed by the U.S. Army Medical Department and the Veterans Health Administration. While progress has been made in PTSD treatment, data from the World Mental Health Survey have recently shown that rates of recovery from combat-related PTSD, world-wide, are approximately one-half the rates of recovery from other trauma types. Furthermore, other recent studies have reported that effect sizes shown by evidence-based treatments for PTSD when applied to male patients are approximately half of what they are when applied to female patients. These results suggest the VA has far to go in achieving efficacious and effective behavioral treatments for this diagnosis affecting a large proportion of its patient population.

In the course of a DoD-funded study (Can a Canine Companion Modify Cardiac Autonomic Reactivity and Tone in PTSD) our laboratory has found that the presence of a service canine in the testing chamber in close proximity to the participant is associated with modification of visual attentional bias away from angry faces signalling social threat along with attenuation of autonomic responses to loud tones. The attenuation of bias towards social threat is of particular relevance to the social impairments seen in this disorder.Veterans with chronic severe PTSD frequently manifest impairments in the execution of key social roles such as those of spouse, parent and employee.

Service canine companionship and oxytocin (OT) appear to be on parallel tracks as novel candidate PTSD treatments or treatment enhancers. A wealth of anecdotal evidence has emerged from U.S. military clinical settings supporting the benefits of service canine companionship and canine-assisted interventions for military personnel with deployment-related mental health conditions; however, rigorously empirical support for this approach remains sparse. A growing literature exploring the role(s) of the OT system in PTSD now includes a number of encouraging findings. For example, in PTSD, OT modulates amygdala hemodynamic responses to emotional faces and increases anterior insula hemodynamic responses to social rewards. Intranasal OT administration normalizes amygdala functional connectivity in PTSD and increased subjective compassion for other persons. These findings align with findings in healthy persons. After intranasal administration, normal adults gaze more at the eye region of faces, have better memory for faces, are better able to infer the mental states of others, have more positive communications, are more generous, rate faces as more trustworthy owe, and exhibit increased trust behavior. OT also attenuates startle in healthy persons, attenuates amygdala responses to fear-inducing stimuli, and inhibits the stress-responsive release of cortisol. In turn, the human findings generally agree with a large animal literature showing that OT plays an important role in social behaviors such as partner preference, social bonding, and social cognition, while OT dysregulation produces a variety of social impairments.

A recent study published in Science showing that urinary OT levels are elevated in association with mutual gaze between dogs and their owners suggests these two lines of research may be converged on the target of PTSD. The investigators will compare the pattern of results of tests of attention bias and startle induced by intranasal OT (vs placebo) to those the investigators have shown to be induced by the presence (vs absence) of a service dog in Veterans diagnosed with PTSD.

Specific Aim 1: To test the effects of a single-dose OT administration in adults with PTSD on the pattern of performance on a set of laboratory tasks which have previously been administered to similar persons who were or were not accompanied by a service canine on separate occasions.

Hypothesis 1: Following single-dose OT administration, participants will exhibit attenuation of attentional bias toward negatively-valenced content, in general, and toward facial cues denoting social threat, in particular.

Hypothesis 2: Following single-dose OT administration, participants will exhibit reduced cardioacceleratory responses to loud tones and attenuated autonomic responses to a math stressor.

Preliminary power calculations indicate that a sample of 40 subjects in this within-subjects design will yield excellent power to detect a medium size effect (Critical t(38) = 2.02, α = .05, 1- β = .90) for the primary attentional bias measures.

ELIGIBILITY:
Inclusion Criteria:

* US military Veteran
* Current posttraumatic stress disorder
* Medically healthy

Exclusion Criteria:

* DSM-5 diagnosis of schizophrenia, schizoaffective disorder, or psychotic disorder
* Active drug or alcohol use disorder within past 90 days
* Currently participating in a clinical drug trial
* Regular nasal obstruction or nosebleeds (use of saline or nasal decongestant permitted if subject has transient cold only)
* Active medical problems: unstable seizures, significant physical illness (e.g., serious liver, renal, or cardiac pathology)
* Sensitivity to preservatives, in particular E 216, E 218, and chlorobutanol hemihydrate
* Significant hearing or vision impairments
* Habitually drinks large volumes of water

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because data obtained by the investigators were exclusively from male combat veterans, and because the inclusion of female veterans presents challenges related to both variable interaction with gonadal hormones over the menstrual cycle and the need to test for pregnancy, only males will be enrolled into this protocol.
Enrollment: 17 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Change in attentional bias | 1-2 weeks
  Changes between oxytocin vs. placebo lab sessions in the asymmetric allocation of visual attention to one or another of a pair of visual stimuli presented simultaneously as quantified by gaze tracking
Change in startle response -heart rate | 1-2 weeks
  Difference between oxytocin vs. placebo lab sessions in the magnitude of pre-to-post startle stimulus change in heart rate

OTHER OUTCOMES:
Change in startle response -EDA | 1-2 weeks
  Difference between oxytocin vs. placebo lab sessions in the magnitude of pre-to-post startle stimulus change in AC-coupled electrodermal activity at the hand
Change in startle response -EMG | 1-2 weeks
  Difference between oxytocin vs. placebo lab sessions in the magnitude of pre-to-post startle stimulus change in corrugator electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Woodward, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagasawa M, Mitsui S, En S, Ohtani N, Ohta M, Sakuma Y, Onaka T, Mogi K, Kikusui T. Social evolution. Oxytocin-gaze positive loop and the coevolution of human-dog bonds. Science. 2015 Apr 17;348(6232):333-6. doi: 10.1126/science.1261022. Epub 2015 Apr 16. PMID 25883356
- [Background] Ayers LW, Missig G, Schulkin J, Rosen JB. Oxytocin reduces background anxiety in a fear-potentiated startle paradigm: peripheral vs central administration. Neuropsychopharmacology. 2011 Nov;36(12):2488-97. doi: 10.1038/npp.2011.138. Epub 2011 Jul 27. PMID 21796104
- [Background] Baumgartner T, Heinrichs M, Vonlanthen A, Fischbacher U, Fehr E. Oxytocin shapes the neural circuitry of trust and trust adaptation in humans. Neuron. 2008 May 22;58(4):639-50. doi: 10.1016/j.neuron.2008.04.009. PMID 18498743
- [Background] Beery AK, Zucker I. Oxytocin and same-sex social behavior in female meadow voles. Neuroscience. 2010 Aug 25;169(2):665-73. doi: 10.1016/j.neuroscience.2010.05.023. Epub 2010 May 16. PMID 20580660
- [Background] Benjet C, Bromet E, Karam EG, Kessler RC, McLaughlin KA, Ruscio AM, Shahly V, Stein DJ, Petukhova M, Hill E, Alonso J, Atwoli L, Bunting B, Bruffaerts R, Caldas-de-Almeida JM, de Girolamo G, Florescu S, Gureje O, Huang Y, Lepine JP, Kawakami N, Kovess-Masfety V, Medina-Mora ME, Navarro-Mateu F, Piazza M, Posada-Villa J, Scott KM, Shalev A, Slade T, ten Have M, Torres Y, Viana MC, Zarkov Z, Koenen KC. The epidemiology of traumatic event exposure worldwide: results from the World Mental Health Survey Consortium. Psychol Med. 2016 Jan;46(2):327-43. doi: 10.1017/S0033291715001981. Epub 2015 Oct 29. PMID 26511595
- [Background] Ditzen B, Schaer M, Gabriel B, Bodenmann G, Ehlert U, Heinrichs M. Intranasal oxytocin increases positive communication and reduces cortisol levels during couple conflict. Biol Psychiatry. 2009 May 1;65(9):728-31. doi: 10.1016/j.biopsych.2008.10.011. Epub 2008 Nov 22. PMID 19027101
- [Background] Domes G, Heinrichs M, Michel A, Berger C, Herpertz SC. Oxytocin improves "mind-reading" in humans. Biol Psychiatry. 2007 Mar 15;61(6):731-3. doi: 10.1016/j.biopsych.2006.07.015. Epub 2006 Nov 29. PMID 17137561
- [Background] Ellenbogen MA, Linnen AM, Cardoso C, Joober R. Intranasal oxytocin attenuates the human acoustic startle response independent of emotional modulation. Psychophysiology. 2014 Nov;51(11):1169-77. doi: 10.1111/psyp.12263. Epub 2014 Aug 1. PMID 25082371
- [Background] Frijling JL, van Zuiden M, Koch SB, Nawijn L, Veltman DJ, Olff M. Effects of intranasal oxytocin on amygdala reactivity to emotional faces in recently trauma-exposed individuals. Soc Cogn Affect Neurosci. 2016 Feb;11(2):327-36. doi: 10.1093/scan/nsv116. Epub 2015 Sep 17. PMID 26382634
- [Background] Guastella AJ, Mitchell PB, Dadds MR. Oxytocin increases gaze to the eye region of human faces. Biol Psychiatry. 2008 Jan 1;63(1):3-5. doi: 10.1016/j.biopsych.2007.06.026. Epub 2007 Sep 21. PMID 17888410
- [Background] Galovski TE, Blain LM, Chappuis C, Fletcher T. Sex differences in recovery from PTSD in male and female interpersonal assault survivors. Behav Res Ther. 2013 Jun;51(6):247-55. doi: 10.1016/j.brat.2013.02.002. Epub 2013 Mar 1. PMID 23510841
- [Background] Kirsch P, Esslinger C, Chen Q, Mier D, Lis S, Siddhanti S, Gruppe H, Mattay VS, Gallhofer B, Meyer-Lindenberg A. Oxytocin modulates neural circuitry for social cognition and fear in humans. J Neurosci. 2005 Dec 7;25(49):11489-93. doi: 10.1523/JNEUROSCI.3984-05.2005. PMID 16339042
- [Background] Koch SB, van Zuiden M, Nawijn L, Frijling JL, Veltman DJ, Olff M. Intranasal Oxytocin Normalizes Amygdala Functional Connectivity in Posttraumatic Stress Disorder. Neuropsychopharmacology. 2016 Jul;41(8):2041-51. doi: 10.1038/npp.2016.1. Epub 2016 Jan 7. PMID 26741286
- [Background] Kosfeld M, Heinrichs M, Zak PJ, Fischbacher U, Fehr E. Oxytocin increases trust in humans. Nature. 2005 Jun 2;435(7042):673-6. doi: 10.1038/nature03701. PMID 15931222
- [Background] Macbeth AH, Stepp JE, Lee HJ, Young WS 3rd, Caldwell HK. Normal maternal behavior, but increased pup mortality, in conditional oxytocin receptor knockout females. Behav Neurosci. 2010 Oct;124(5):677-85. doi: 10.1037/a0020799. PMID 20939667
- [Background] Nawijn L, van Zuiden M, Koch SB, Frijling JL, Veltman DJ, Olff M. Intranasal oxytocin increases neural responses to social reward in post-traumatic stress disorder. Soc Cogn Affect Neurosci. 2017 Feb 1;12(2):212-223. doi: 10.1093/scan/nsw123. PMID 27614769
- [Background] Palgi S, Klein E, Shamay-Tsoory SG. Oxytocin improves compassion toward women among patients with PTSD. Psychoneuroendocrinology. 2016 Feb;64:143-9. doi: 10.1016/j.psyneuen.2015.11.008. Epub 2015 Nov 17. PMID 26671007
- [Background] Rimmele U, Hediger K, Heinrichs M, Klaver P. Oxytocin makes a face in memory familiar. J Neurosci. 2009 Jan 7;29(1):38-42. doi: 10.1523/JNEUROSCI.4260-08.2009. PMID 19129382
- [Background] Rubenstein DA, Debboun M, Burton R. Canine-assisted therapy in military medicine. Perspectives: commander's introduction. US Army Med Dep J. 2012 Apr-Jun:1-4. No abstract available. PMID 22512055
- [Background] Theodoridou A, Rowe AC, Penton-Voak IS, Rogers PJ. Oxytocin and social perception: oxytocin increases perceived facial trustworthiness and attractiveness. Horm Behav. 2009 Jun;56(1):128-32. doi: 10.1016/j.yhbeh.2009.03.019. Epub 2009 Apr 1. PMID 19344725
- [Background] Wade D, Varker T, Kartal D, Hetrick S, O'Donnell M, Forbes D. Gender difference in outcomes following trauma-focused interventions for posttraumatic stress disorder: Systematic review and meta-analysis. Psychol Trauma. 2016 May;8(3):356-64. doi: 10.1037/tra0000110. Epub 2016 Feb 8. PMID 26854354
- [Background] Zak PJ, Stanton AA, Ahmadi S. Oxytocin increases generosity in humans. PLoS One. 2007 Nov 7;2(11):e1128. doi: 10.1371/journal.pone.0001128. PMID 17987115